CLINICAL TRIAL: NCT04521478
Title: A Phase II, 6-week, Multicenter, Randomized, Double-blind, Double-dummy, Placebo-controlled, Parallel Group Trial With a Quetiapine Arm to Evaluate the Efficacy, Tolerability and Safety of Oral BI 1358894 in Patients With Major Depressive Disorder With Inadequate Response to Antidepressants.
Brief Title: A Study to Test the Effect of Different Doses of BI 1358894 and Quetiapine in People With Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1402-0011; 2019-004264-21 (EudraCT Number)
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — TRPC inhibitor BI 1358894; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 5 mg BI 1358894 (Experimental): Participants with an established diagnosis of MDD administered one 5 milligram (mg) dose of BI 1358894 in the morning as film-coated tablet, and one dose of placebo matching quetiapine in the evening as tablets. Each administration was performed orally once daily, for 6 weeks.
  During the trial, participants also continued treatment with their OAD.
  Interventions: Drug: BI 1358894
- Placebo (Placebo Comparator): Participants with an established diagnosis of Major Depressive Disorder (MDD) administered one dose of placebo matching BI 1358894 in the morning as film-coated tablets, and one dose of placebo matching quetiapine in the evening as tablets. Each administration was performed orally once daily, for 6 weeks.
  During the trial, participants also continued treatment with their Ongoing Antidepressants (OAD).
  Interventions: Drug: Placebo
- Quetiapine (Active Comparator): Participants with an established diagnosis of MDD administered one dose of placebo matching BI 1358894 in the morning as film-coated tablets, and one 150 or 300 mg dose of quetiapine in the evening as tablets. Each administration was performed orally once daily, for 6 weeks.
  The daily active dose at the start of therapy was 50 mg on Day 1, 100 mg at Day 2 and 150 mg on Day 3 and 4. Beginning with Day 5, the recommended daily dose of 300 mg was taken. If not tolerated by a participant, the dose was reduced to 150 mg in Week 1. Thereafter, this finally chosen dose had to be stable until end of treatment at Week 6.
  During the trial, participants also continued treatment with their OAD.
  Interventions: Drug: Quetiapine
- 25 mg BI 1358894 (Experimental): Participants with an established diagnosis of MDD administered one 25 mg dose of BI 1358894 in the morning as film-coated tablet, and one dose of placebo matching quetiapine in the evening as tablets. Each administration was performed orally once daily, for 6 weeks.
  During the trial, participants also continued treatment with their OAD.
  Interventions: Drug: BI 1358894
- 75 mg BI 1358894 (Experimental): Participants with an established diagnosis of MDD administered one 75 mg dose of BI 1358894 in the morning as film-coated tablets, and one dose of placebo matching quetiapine in the evening as tablets. Each administration was performed orally once daily, for 6 weeks.
  During the trial, participants also continued treatment with their OAD.
  Interventions: Drug: BI 1358894
- 125 mg BI 1358894 (Experimental): Participants with an established diagnosis of MDD administered one 125 mg dose of BI 1358894 in the morning as film-coated tablets, and one dose of placebo matching quetiapine in the evening as tablets. Each administration was performed orally once daily, for 6 weeks.
  During the trial, participants also continued treatment with their OAD.
  Interventions: Drug: BI 1358894

INTERVENTIONS:
Drug: BI 1358894 — BI 1358894
  Arms: 125 mg BI 1358894; 25 mg BI 1358894; 5 mg BI 1358894; 75 mg BI 1358894
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Quetiapine — quetiapine
  Arms: Quetiapine

SUMMARY:
This study is open to adults with depression (major depressive disorder) for whom standard treatment with antidepressants alone does not work sufficiently. The purpose of the trial is to find out whether a medicine called BI 1358894 helps to improve symptoms of depression. Four different doses of BI 1358894 are tested in the study. Participants continue their standard antidepressant therapy throughout the study. Participants are put into 6 groups by chance. Participants in 4 of the 6 groups take different doses of BI 1358894, and placebo. Participants in the fifth group take quetiapine, a medicine already used to treat depression, and placebo. Participants in the sixth group take placebo only.

Participants take BI 1358894, quetiapine, or placebo as tablets. Placebo tablets look like BI 1358894 or quetiapine tablets but do not contain any medicine. Each participant takes tablets twice a day. Participants are in the study for about 3 months. During this time, they visit the study site about 8 times and get about 2 phone calls. At the visits, doctors ask participants about their symptoms.

The results between the BI 1358894 groups, the quetiapine group, and the placebo group are then compared. The doctors also regularly check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

--Established diagnosis of Major Depressive Disorder (MDD), single episode or recurrent, as confirmed at the time of screening by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, 5th version (DSM-5) (SCID-5), with a duration of current depressive episode ≥ 8 weeks and ≤ 24 months at the time of screening visit

* Montgomery-Åsberg Depression Rating Scale (MADRS) total score ≥ 24 at screening, as confirmed by a trained site based rater AND interactive, computer administered MADRS. The difference in the rater and computer administered MADRS must not exceed more than 7 points (for details refer to section 6.2). In addition, trial participants must have a score of ≥ 3 on the Reported Sadness Item on both MADRS scales (computer administered and rater-administered MADRS)
* A documented ongoing monotherapy treatment of ≥ 4 weeks at the screening visit, with bupropion or a protocol specified Selective Serotonin Reuptake Inhibitor (SSRI) or Serotonin Norepinephrine Reuptake Inhibitor (SNRI) (refer to the ISF) at adequate dose (at least minimum effective dose as per prescribing information and as confirmed per detectable drug levels in the screening blood or urine sampling)
* Male and female participants, 18 to 65 years of age, both inclusively at the time of consent
* Women who are of child-bearing potential (WOCBP)1 must be able and willing, as confirmed by the investigator, to use two methods of contraception which include one highly effective method of birth control per ICH M3 (R2) that result in a low failure rate of less than 1%, plus one additional barrier
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
* Able to communicate well, and to understand and comply with trial requirements

Exclusion Criteria:

* Per DSM-5, had ever met diagnostic criteria for schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar disorder, delusional disorder or MDD with psychotic features as assessed by the Structured Clinical Interview for DSM-5 Clinical Trials (SCID-5) at the time of screening
* Diagnosis of any other mental disorder (in addition to those as described in Exclusion Criterion #1) that was the primary focus of treatment within 6 months prior to screening or at baseline (as per clinical discretion of the investigator)
* Diagnosis with antisocial, paranoid, schizoid or schizotypal personality disorder as per DSM-5 criteria, at the time of screening visit. Any other personality disorder at screening visit that significantly affects current psychiatric status and likely to impact trial participation, as per the judgement of investigator
* Diagnosis of a substance related disorder within 3 months prior to screening visit (with exception of caffeine and tobacco)
* History of seizure disorders, stroke, brain tumor or any other major neurological illness that can impact participation in the trial
* History of more than 2 unsuccessful monotherapy treatments (at adequate dosage and duration, per local prescribing information of the product) with an approved antidepressant medication for the current ongoing major depressive episode. These include ongoing monotherapy treatment with bupropion or a protocol specified SSRI or SNRI as described in Inclusion Criterion #3
* Any suicidal behavior in the past 12 months prior to screening (per investigator judgement including an actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behaviour)
* Any suicidal ideation of type 4 or 5 in the Columbia Suicide Severity Rating Scale (CSSRS) in the past 3 months prior to screening or at screening or baseline visit (i.e. active suicidal thought with method and intent but without specific plan, or active suicidal thought with method, intent and plan)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-02-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (120):
- United States (29):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Collaborative Neuroscience Network, LLC (CNS), Garden Grove, California
  - Alliance Research, Long Beach, California
  - Asclepes Research Centers, Sherman Oaks, California
  - California Neuroscience Research, Sherman Oaks, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Viking Clinical Research, Ltd., Temecula, California
  - Collaborative Neuroscience Research, LLC, Torrance, California
  - Mountain Mind. LLC, Denver, Colorado
  - CT Clinical Research, Cromwell, Connecticut
  - Institute of Living, Hartford, Connecticut
  - Gulf Coast Clinical Research Center, Fort Myers, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Optimus U Corporation, Miami, Florida
  - Advanced Discovery Research LLC, Atlanta, Georgia
  - Atlanta Center, Atlanta, Georgia
  - Chicago Research Center, Incorporated, Chicago, Illinois
  - University of Kansas School of Medicine-Wichita, Wichita, Kansas
  - Precise Research Centers, Flowood, Mississippi
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - Center For Emotional Fitness, Cherry Hill, New Jersey
  - Hassman Research Institute, Marlton, New Jersey
  - Synexus Clinical Research US, Inc., New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Global Medical Institutes, LLC, Scranton Medical Institute, Moosic, Pennsylvania
  - Core Clinical Research, Everett, Washington
- Argentina (8):
  - Fundación para el Estudio y Tratamiento de las Enfermedades Mentales (FETEM), CABA
  - CEN (Centro Especializado Neurociencias), Córdoba
  - Instituto DAMIC - Fundacion Rusculleda, Córdoba
  - CENPIA-Centro de Estudios Neuropsiquiátricos y Psicológicos Integral Ambulatorio, La Plata
  - Clinica Privada de Salud Mental Santa Teresa de Avila, La Plata
  - Instituto de Neurociencias San Agustín, La Plata
  - Instituto Médico de la Fundación Estudios Clínicos, Rosario
  - Centro de Investigacion y Asistencia en Psiquiatria (CIAP), Rosario
- Australia (4):
  - Griffith Health, Southport, Queensland
  - Peninsula Therapeutic and Research Group, Frankston, Victoria
  - Albert Road Clinic, Melbourne, Victoria
  - Monash Alfred Psychiatry Research Centre, Melbourne, Victoria
- Bulgaria (3):
  - Mental Health Center "Prof. Dr. Ivan Temkov - Burgas" EOOD, Burgas
  - Filipopolis Ambulatory for Group Practice for Specialized Care in Psychiatry, Plovdiv
  - Medical Center Intermedica Ltd., Sofia
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - OCT Research ULC, Kelowna, British Columbia
  - Braxia Scientific Corp. (CRTCE Mississauga), Mississauga, Ontario
  - Centre for Addiction and Mental Health (CAMH), Toronto, Ontario
- Czechia (7):
  - Neuropsychiatry, s.r.o., Hradec Králové
  - Clinical Research Foundation s.r.o, Kladno
  - MP Meditrine s.r.o., Ostrava
  - A-SHINE s.r.o, Pilsen
  - Clintrial s.r.o., Prague
  - AD71 s.r.o., Prague
  - INEP medical s.r.o., Prague
- France (9):
  - HOP Dijon-Bourgogne, Dijon
  - CAB Médical Psyché, Douai
  - CAB Ambroise Paré, Élancourt
  - HOP la Colombière, Montpellier
  - HOP Saint-Jacques, Nantes
  - HOP Pasteur, Nice
  - HOP Carémeau, Nîmes
  - CTR Psychiatrique Universitaire, Saint-Cyr-sur-Loire
  - HOP Purpan, Toulouse
- Germany (6):
  - Zentrum für klinische Forschung Dr. med. I. Schöll GmbH, Bad Homburg
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Zentralinstitut für seelische Gesundheit, Mannheim
  - Praxis für Psychiatrie und Psychotherapie, Stralsund
  - Studienzentrum Nord-West, Westerstede
- Hungary (3):
  - Obuda Health Center, Budapest
  - Semmelweis University, Budapest
  - Bugat Pal Hospital, Gyongyos, Gyöngyös
- Japan (20):
  - National Center for Global Health and Medicine Kohnodai Hospital, Chiba, Ichikawa
  - Kaku Mental Clinic, Fukuoka, Fukuoka
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Kuramitsu Hospital, Fukuoka, Fukuoka
  - Hokudai-dori Mental Health Clinic, Hokkaido, Sapporo
  - Arai Clinic, Hyogo, Amagasaki
  - Tatsuta Clinic, Hyogo, Kobe
  - Kishiro Mental Clinic, Kanagawa, Kawasaki
  - Yutaka Clinic, Kanagawa,Sagamihara
  - Yuge Neuropsychiatric Hospital, Kumamoto, Kumamoto
  - Arata Clinic, Nagasaki, Nagasaki
  - Nara Medical University Hospital, Nara, Kashihara
  - Rainbow and Sea Hospital, Saga, Karatsu
  - Inuo Hospital, Saga, Tosu
  - National Center of Neurology and Psychiatry, Tokyo, Kodaira
  - Tamachi mita cocoromi Clinic, Tokyo, Minato-ku
  - Sancha Mental Clinic, Tokyo, Setagaya-ku
  - Maynds Tower Mental Clinic, Tokyo, Shibuya-ku
  - Ichigaya Himorogi Clinic, Tokyo, Shinjuku-ku
  - Ohwa Mental Clinic, Tokyo, Toshima-ku
- Poland (6):
  - Synexus Polska SCM Sp. z o.o. Gdansku, Gdansk, Gdansk
  - Synexus Lodz Medical Center, Lodz
  - Specialist Psychiatric Healthcare Centre in Lodz, Lodz
  - Clinical Best Solutions, Lublin
  - Centrum Medyczne "Luxmed" Sp. z o.o., Lublin
  - Synexus Poland, Branch in Poznan, Poznan
- Russia (7):
  - Federal State Budget Institution "Mental Health Research Center", Moscow
  - SBI of HC "Z. P. Solovyov Scientific&pract psychoneurolog.Cent", Moscow
  - SBHI "Psychiatric Hospital #1 P.P.Kashchenko", Saint Petersburg
  - FSBI Bekhterev Net.Med.Res.Cen.of Psych&Neuro, Saint Petersburg
  - LLC "MK-Med", Saint Petersburg
  - SHI "Reg.Clin.Psychiatric Hosp.of Saint Sophia", Saratov
  - FSBEI of HE Smolensk State Medical University, Smolensk
- Slovakia (8):
  - MUDr. Beata Dupejová, Banská Bystrica
  - J & J SMART, s.r.o., psychiatric clinic, Bratislava
  - MENTUM s.r.o., Bratislava
  - EPAMED s.r.o., Košice
  - Psychiatricka klinika I.UN L. Pasteura, Košice
  - CENTRUM ZDRAVIA R.B.K, s.r.o., psychiatric clinic, Svidník
  - Pro mente sana s.r.o., Psychiatric clinic, Trenčín
  - Crystal Comfort s.r.o, Vranov nad Topľou
- Spain (6):
  - Hospital Universitario Fundación Alcorcón, Alcorcón
  - Hestia Palau, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Jerez de la Frontera, Jerez de la Frontera
  - Hospital Ramón y Cajal, Madrid
  - Centro de Salud de San Juan, Salamanca

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Shelton RC, Pizzagalli DA, Cohen EA, Hori H, Dickschat U, Asafu-Adjei J, Feldbarg A, Just S, Roehrle M, Sommer S, Sussmuth SD. Efficacy, Tolerability, and Safety of TRPC4/5 Inhibitor BI 1358894 in Patients With Major Depressive Disorder and Inadequate Response to Antidepressants: A Phase 2 Randomized, Placebo-Controlled, Parallel Group, Dose-Ranging Trial. J Clin Psychiatry. 2025 Sep 3;86(3):25m15868. doi: 10.4088/JCP.25m15868. PMID 40900110
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase II, 6-week parallel-group multicenter, randomized, double blind, doubledummy, placebo-controlled trial with a Quetiapine arm in participants with Major Depressive Disorder (MDD) with inadequate response to ongoing treatment with a Selective Serotonin Reuptake Inhibitor (SSRI) or a Serotonin Norepinephrine Reuptake Inhibitor (SNRI) or bupropion.
Pre-assignment Details: All patients were screened for eligibility prior to participation in the trial, to ensure that they met all inclusion and none of the exclusion criteria.
  One patient was randomized to the placebo arm but treated with 125 mg BI 1358894.
Period: Overall Study
Arm/Group | Placebo | 5 mg BI 1358894 | 25 mg BI 1358894 | 75 mg BI 1358894 | 125 mg BI 1358894 | Quetiapine
Started | 129 | 36 | 39 | 39 | 74 | 72
Treated (one participant from the "Placebo" arm was treated with 125 mg BI 1358894, and thus was analyzed as part of the "125 mg BI 1358894" arm for the Safety Analyses. This patient is shown here in the "Placebo" arm.) | 129 | 36 | 39 | 39 | 74 | 71
Completed | 116 | 31 | 33 | 34 | 67 | 59
Not Completed | 13 | 5 | 6 | 5 | 7 | 13
Not completed — Protocol Violation | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Technical Problems | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Burden of Study Procedures | 1 | 0 | 0 | 1 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 7 | 0 | 2 | 1 | 2 | 7
Not completed — No Reason Available | 0 | 2 | 0 | 0 | 1 | 0
Not completed — Other than listed | 3 | 3 | 3 | 2 | 3 | 3
Not completed — Not treated | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): all participants that have been randomized and that received at least one administration of study drug. Participants are analysed according to the actual received treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 5 mg BI 1358894 | 25 mg BI 1358894 | 75 mg BI 1358894 | 125 mg BI 1358894 | Quetiapine | Total
Number analyzed (Participants) | 128 | 36 | 39 | 39 | 75 | 71 | 388
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.9 (13.0) | 39.7 (13.8) | 44.7 (12.1) | 42.7 (12.2) | 47.7 (11.7) | 43.6 (12.4) | 43.8 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 27 | 28 | 26 | 51 | 49 | 263
  Male | 46 | 9 | 11 | 13 | 24 | 22 | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 5 | 2 | 5 | 8 | 12 | 51
  Not Hispanic or Latino | 109 | 31 | 37 | 34 | 67 | 59 | 337
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 24 | 5 | 6 | 6 | 15 | 12 | 68
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 2 | 3 | 1 | 7 | 6 | 25
  White | 98 | 29 | 30 | 32 | 53 | 53 | 295
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Montgomery-Åsberg Depression Rating Scale (MADRS) total score [Mean (Standard Deviation); unit: Score on a scale] — The MADRS evaluates core symptoms of depression and consists of 10 items. Nine of them are based upon participant reports, and one is on the rater's observation (apparent sadness) during the rating interview. MADRS items are rated on a 0-6 continuum (0=no abnormality, 6=severe). The possible total score could range from 0 (normal with absence of symptoms) to 60 (severe depression).
  Baseline MADRS total score is the last non-missing value recorded prior to first dose of trial medication.
  Score on a scale | 32.0 (6.4) | 34.0 (4.8) | 34.1 (5.6) | 32.1 (6.4) | 33.1 (6.0) | 33.6 (5.6) | 32.9 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score at Week 6
Description: Change from baseline in MADRS total score at Week 6 is reported. The MADRS evaluates core symptoms of depression and consists of 10 items. Nine of them are based upon participant reports, and one is on the rater's observation (apparent sadness) during the rating interview. MADRS items are rated on a 0-6 continuum (0=no abnormality, 6=severe). The possible total score could range from 0 (normal with absence of symptoms) to 60 (severe depression).
  Least squares mean and adjusted standard error were estimated by Restricted Maximum Likelihood (REML)-based Mixed effects model for repeated measures (MMRM) including the fixed categorical effects of treatment, concomitant psychotherapy use (yes vs. no), and the fixed continuous effect of baseline MADRS total score. Visit was treated as a repeated measure with an unstructured covariance matrix. The Kenward-Roger approximation was used to estimate the denominator degrees of freedom and adjust standard errors.
Time Frame: MMRM included measurements from baseline (Week 0) and at Weeks 1, 2, 4 and 6 after first drug administration. MMRM estimates of change from baseline to Week 6 is reported.
Population: Full analysis set (FAS): all participants in TS that have a baseline and at least one evaluable post-baseline measurement. As per protocol, data from participants assigned to the quetiapine arm were not included in the primary endpoint.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 5 mg BI 1358894 | 25 mg BI 1358894 | 75 mg BI 1358894 | 125 mg BI 1358894
Number analyzed (Participants) | 126 | 36 | 39 | 39 | 72
Units on a scale | -13.0 (1.0) | -12.4 (2.0) | -10.8 (1.9) | -10.8 (1.9) | -11.5 (1.4)
Statistical Analysis 1: Comparison: Placebo vs 5 mg BI 1358894; Adjusted means and confidence intervals were estimated using REML-based MMRM including the fixed categorical effects of treatment, concomitant psychotherapy use (yes vs. no), and the fixed continuous effect of baseline MADRS total score. Visit was treated as a repeated measure with an unstructured covariance matrix. The Kenward-Roger approximation was used to estimate the denominator degrees of freedom and adjust standard errors; Test type: Other; p = 0.7636, Mixed Models Analysis; Mean Difference (Net) = 0.7, 90% CI 2-sided [-3.0 to 4.3], Standard Error of Mean 2.2 — Difference = (adjusted mean 5 mg BI 1358894) - (adjusted mean Placebo)
Statistical Analysis 2: Comparison: Placebo vs 25 mg BI 1358894; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.3040, Mixed Models Analysis; Mean Difference (Net) = 2.3, 90% CI 2-sided [-1.4 to 5.9], Standard Error of Mean 2.2 — Difference = (adjusted mean 25 mg BI 1358894) - (adjusted mean Placebo)
Statistical Analysis 3: Comparison: Placebo vs 75 mg BI 1358894; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.3090, Mixed Models Analysis; Mean Difference (Net) = 2.2, 90% CI 2-sided [-1.4 to 5.7], Standard Error of Mean 2.2 — Difference = (adjusted mean 75 mg BI 1358894) - (adjusted mean Placebo)
Statistical Analysis 4: Comparison: Placebo vs 125 mg BI 1358894; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.3694, Mixed Models Analysis; Mean Difference (Net) = 1.5, 90% CI 2-sided [-1.3 to 4.4], Standard Error of Mean 1.7 — Difference = (adjusted mean 125 mg BI 1358894) - (adjusted mean Placebo)
Statistical Analysis 5: Comparison: Placebo vs 5 mg BI 1358894 vs 25 mg BI 1358894 vs 75 mg BI 1358894 vs 125 mg BI 1358894; The Multiple Comparison Procedures and Modeling (MCPMod) procedure used the estimated values from an MMRM model as input and allowed for simultaneous evaluation of different potential dose response patterns (Linear, Exponential, Emax1, Emax2, Sigmoid Emax), while protecting the overall false positive rate (probability of Type I error) using a one-sided, nominal α level of 10 %; Test type: Other; p = 0.9158, MCPMod Linear model; No parameter assumptions required. Corresponding dose response is linear
Statistical Analysis 6: Comparison: Placebo vs 5 mg BI 1358894 vs 25 mg BI 1358894 vs 75 mg BI 1358894 vs 125 mg BI 1358894; [analysis description as in outcome 1, analysis 5]; Test type: Other; p = 0.8676, MCPMod Exponential model; Assumption: 5% of the maximum effect is achieved at 25 mg; corresponding to a drug effect achieved mainly at higher doses
Statistical Analysis 7: Comparison: Placebo vs 5 mg BI 1358894 vs 25 mg BI 1358894 vs 75 mg BI 1358894 vs 125 mg BI 1358894; [analysis description as in outcome 1, analysis 5]; Test type: Other; p = 0.9552, MCPMod Emax1 model; Assumption: 50% of the maximum effect is achieved at 25 mg; corresponding to the assumed true median effective dose (ED50) = 25 mg
Statistical Analysis 8: Comparison: Placebo vs 5 mg BI 1358894 vs 25 mg BI 1358894 vs 75 mg BI 1358894 vs 125 mg BI 1358894; [analysis description as in outcome 1, analysis 5]; Test type: Other; p = 0.9619, MCPMod Emax2 model; Assumption: 70% of the maximum effect is achieved at 5 mg; corresponding to a drug effect achieved mainly with low doses, ED50 = 2.14 mg
Statistical Analysis 9: Comparison: Placebo vs 5 mg BI 1358894 vs 25 mg BI 1358894 vs 75 mg BI 1358894 vs 125 mg BI 1358894; [analysis description as in outcome 1, analysis 5]; Test type: Other; p = 0.9507, MCPMod Sigmoid Emax model; Assumption: 50% of the maximum effect is achieved at 25 mg, 90% 75 mg; corresponding to a more flexible model of the assumed true ED50 = 25 mg

2. Secondary Outcome: Number of Participants With Response Defined as ≥ 50% Montgomery-Åsberg Depression Rating Scale (MADRS) Reduction From Baseline at Week 6
Description: Number of participants with response defined as ≥ 50% MADRS reduction from baseline at Week 6 is reported. Percent reduction from baseline was calculated as follows: [(MADRS total score at baseline - MADRS total score at week 6)/ MADRS total score at baseline] *100.
Time Frame: Prior to the first intake of the trial medication (week 0, baseline) and after 6 weeks of treatment.
Population: Full analysis set (FAS): all participants in TS that have a baseline and at least one evaluable post-baseline measurement. As per protocol, data from participants assigned to the quetiapine arm were not included in the secondary endpoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 5 mg BI 1358894 | 25 mg BI 1358894 | 75 mg BI 1358894 | 125 mg BI 1358894
Number analyzed (Participants) | 126 | 36 | 39 | 39 | 72
Participants | 40 | 10 | 9 | 12 | 23
Statistical Analysis 1: Comparison: Placebo vs 5 mg BI 1358894; Logistic regression model, including the fixed categorical effects of treatment and baseline MDD severity; Test type: Other; p = 0.8889, Regression, Logistic; Odds Ratio (OR) = 0.9427, 90% CI 2-sided [0.4709 to 1.8873] — 5 mg BI 1358894 vs Placebo
Statistical Analysis 2: Comparison: Placebo vs 25 mg BI 1358894; Logistic regression model, including the fixed categorical effects of treatment and baseline MDD severity; Test type: Other; p = 0.3284, Regression, Logistic; Odds Ratio (OR) = 0.6581, 90% CI 2-sided [0.3255 to 1.3307] — 25 mg BI 1358894 vs Placebo
Statistical Analysis 3: Comparison: Placebo vs 75 mg BI 1358894; Logistic regression model, including the fixed categorical effects of treatment and baseline MDD severity; Test type: Other; p = 0.8048, Regression, Logistic; Odds Ratio (OR) = 1.1026, 90% CI 2-sided [0.5757 to 2.1114] — 75 mg BI 1358894 vs Placebo
Statistical Analysis 4: Comparison: Placebo vs 125 mg BI 1358894; Logistic regression model, including the fixed categorical effects of treatment and baseline MDD severity; Test type: Other; p = 0.9820, Regression, Logistic; Odds Ratio (OR) = 1.0072, 90% CI 2-sided [0.5968 to 1.6999] — 125 mg BI 1358894 vs Placebo

3. Secondary Outcome: Change From Baseline in State-Trait Anxiety Inventory (STAI) State and Trait Version Scores at Week 6
Description: Change from baseline in STAI State and Trait version scores at Week 6 is reported. The STAI comprises separate self-report scales for measuring state and trait anxiety. Both consist of 20 statements. The S-Anxiety scale evaluates how respondents feel "right now, at this moment." The T-Anxiety scale assesses how people generally feel. Each STAI item is given a weighted score of 1 to 4. Scores for both scales can vary from 20 (minimum) to 80 (maximum). Higher scores indicate greater anxiety.
  Least squares mean and adjusted standard error were estimated by REML-based MMRM including the fixed categorical effects of treatment, concomitant psychotherapy use (yes vs. no), and the fixed continuous effect of baseline score. Visit was treated as a repeated measure with an unstructured covariance matrix. The Kenward-Roger approximation was used to estimate the denominator degrees of freedom and adjust standard errors.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 5 mg BI 1358894 | 25 mg BI 1358894 | 75 mg BI 1358894 | 125 mg BI 1358894
Number analyzed (Participants) | 126 | 36 | 39 | 39 | 72
Units on a scale
  S-Anxiety | -11.3 (1.2) | -7.0 (2.3) | -8.9 (2.3) | -12.3 (2.2) | -8.6 (1.6)
  T-Anxiety | -11.0 (1.1) | -6.9 (2.1) | -10.2 (2.1) | -9.9 (2.1) | -7.2 (1.5)
Statistical Analysis 1: Comparison: Placebo vs 5 mg BI 1358894; Adjusted means and confidence intervals were estimated using REML-based MMRM including the fixed categorical effects of treatment, concomitant psychotherapy use (yes vs. no), and the fixed continuous effect of baseline score (S-Anxiety scale). Visit was treated as a repeated measure with an unstructured covariance matrix. The Kenward-Roger approximation was used to estimate the denominator degrees of freedom and adjust standard errors; Test type: Other; p = 0.1013, Mixed Models Analysis; Mean Difference (Net) = 4.3, 90% CI 2-sided [0.0 to 8.6], Standard Error of Mean 2.6 — Difference = (adjusted mean 5 mg BI 1358894) - (adjusted mean Placebo)
Statistical Analysis 2: Comparison: Placebo vs 25 mg BI 1358894; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.3596, Mixed Models Analysis; Mean Difference (Net) = 2.4, 90% CI 2-sided [-1.9 to 6.6], Standard Error of Mean 2.6 — Difference = (adjusted mean 25 mg BI 1358894) - (adjusted mean Placebo)
Statistical Analysis 3: Comparison: Placebo vs 75 mg BI 1358894; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.6745, Mixed Models Analysis; Mean Difference (Net) = -1.1, 90% CI 2-sided [-5.2 to 3.1], Standard Error of Mean 2.5 — Difference = (adjusted mean 75 mg BI 1358894) - (adjusted mean Placebo)
Statistical Analysis 4: Comparison: Placebo vs 125 mg BI 1358894; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.1870, Mixed Models Analysis; Mean Difference (Net) = 2.7, 90% CI 2-sided [-0.7 to 6.0], Standard Error of Mean 2.0 — Difference = (adjusted mean 125 mg BI 1358894) - (adjusted mean Placebo)
Statistical Analysis 5: Comparison: Placebo vs 5 mg BI 1358894; Adjusted means and confidence intervals were estimated using REML-based MMRM including the fixed categorical effects of treatment, concomitant psychotherapy use (yes vs. no), and the fixed continuous effect of baseline score (T-Anxiety scale). Visit was treated as a repeated measure with an unstructured covariance matrix. The Kenward-Roger approximation was used to estimate the denominator degrees of freedom and adjust standard errors; Test type: Other; p = 0.0921, Mixed Models Analysis; Mean Difference (Net) = 4.1, 90% CI 2-sided [0.1 to 8.1], Standard Error of Mean 2.4 — Difference = (adjusted mean 5 mg BI 1358894) - (adjusted mean Placebo)
Statistical Analysis 6: Comparison: Placebo vs 25 mg BI 1358894; [analysis description as in outcome 3, analysis 5]; Test type: Other; p = 0.7395, Mixed Models Analysis; Mean Difference (Net) = 0.8, 90% CI 2-sided [-3.2 to 4.8], Standard Error of Mean 2.4 — Difference = (adjusted mean 25 mg BI 1358894) - (adjusted mean Placebo)
Statistical Analysis 7: Comparison: Placebo vs 75 mg BI 1358894; [analysis description as in outcome 3, analysis 5]; Test type: Other; p = 0.6296, Mixed Models Analysis; Mean Difference (Net) = 1.1, 90% CI 2-sided [-2.7 to 5.0], Standard Error of Mean 2.4 — Difference = (adjusted mean 75 mg BI 1358894) - (adjusted mean Placebo)
Statistical Analysis 8: Comparison: Placebo vs 125 mg BI 1358894; [analysis description as in outcome 3, analysis 5]; Test type: Other; p = 0.0429, Mixed Models Analysis; Mean Difference (Net) = 3.8, 90% CI 2-sided [0.7 to 6.9], Standard Error of Mean 1.9 — Difference = (adjusted mean 125 mg BI 1358894) - (adjusted mean Placebo)

4. Secondary Outcome: Change From Baseline in Clinical Global Impression Severity Scale (CGI-S) Score at Week 6
Description: Change from baseline in CGI-S score at Week 6 is reported. The CGI-S rating scale evaluates the severity of psychopathology on a scale of 1 to 7. Considering total clinical experience with the depression population, a participant is assessed on severity of illness at the time of rating according to: 1=normal (not at all ill); 2=borderline ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill participants.
  Least squares mean and adjusted standard error were estimated by REML-based MMRM including the fixed categorical effects of treatment, concomitant psychotherapy use (yes vs. no), and the fixed continuous effect of the baseline score. Visit was treated as a repeated measure with an unstructured covariance matrix. The Kenward-Roger approximation was used to estimate the denominator degrees of freedom and adjust standard errors.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 5 mg BI 1358894 | 25 mg BI 1358894 | 75 mg BI 1358894 | 125 mg BI 1358894
Number analyzed (Participants) | 126 | 36 | 39 | 39 | 72
Units on a scale | -1.3 (0.1) | -1.2 (0.2) | -1.2 (0.2) | -1.1 (0.2) | -1.1 (0.2)
Statistical Analysis 1: Comparison: Placebo vs 5 mg BI 1358894; Adjusted means and confidence intervals were estimated using REML-based MMRM including the fixed categorical effects of treatment, concomitant psychotherapy use (yes vs. no), and the fixed continuous effect of the baseline score. Visit was treated as a repeated measure with an unstructured covariance matrix. The Kenward-Roger approximation was used to estimate the denominator degrees of freedom and adjust standard errors; Test type: Other; p = 0.6211, Mixed Models Analysis; Mean Difference (Net) = 0.1, 90% CI 2-sided [-0.3 to 0.5], Standard Error of Mean 0.3 — Difference = (adjusted mean 5 mg BI 1358894) - (adjusted mean Placebo)
Statistical Analysis 2: Comparison: Placebo vs 25 mg BI 1358894; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.5158, Mixed Models Analysis; Mean Difference (Net) = 0.2, 90% CI 2-sided [-0.2 to 0.6], Standard Error of Mean 0.2 — Difference = (adjusted mean 25 mg BI 1358894) - (adjusted mean Placebo)
Statistical Analysis 3: Comparison: Placebo vs 75 mg BI 1358894; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.4518, Mixed Models Analysis; Mean Difference (Net) = 0.2, 90% CI 2-sided [-0.2 to 0.6], Standard Error of Mean 0.2 — Difference = (adjusted mean 75 mg BI 1358894) - (adjusted mean Placebo)
Statistical Analysis 4: Comparison: Placebo vs 125 mg BI 1358894; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.2347, Mixed Models Analysis; Mean Difference (Net) = 0.2, 90% CI 2-sided [-0.1 to 0.6], Standard Error of Mean 0.2 — Difference = (adjusted mean 125 mg BI 1358894) - (adjusted mean Placebo)

5. Secondary Outcome: Change From Baseline in Symptoms of Major Depressive Disorder Scale (SMDDS) Total Score at Week 6
Description: Change from baseline in SMDDS total score at Week 6 is reported. The SMDDS is a 16-item, patient-reported outcome measure developed to capture the core symptoms of MDD. The SMDDS uses a recall of "over the past 7 days" and participants respond to each question using a rating scale between 0 ("Not at all" or "Never") to 4 ("Extremely" or "Always"). The total score ranges from 0 to 60 with a higher score indicating more severe depressive symptomatology.
  Least squares mean and adjusted standard error were estimated by REML-based MMRM including the fixed categorical effects of treatment, concomitant psychotherapy use (yes vs. no), and the fixed continuous effect of the baseline score. Visit was treated as a repeated measure with an unstructured covariance matrix. The Kenward-Roger approximation was used to estimate the denominator degrees of freedom and adjust standard errors.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 5 mg BI 1358894 | 25 mg BI 1358894 | 75 mg BI 1358894 | 125 mg BI 1358894
Number analyzed (Participants) | 126 | 36 | 39 | 39 | 72
Units on a scale | -13.3 (1.2) | -9.9 (2.2) | -8.9 (2.2) | -12.3 (2.1) | -10.5 (1.6)
Statistical Analysis 1: Comparison: Placebo vs 5 mg BI 1358894; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.1723, Mixed Models Analysis; Mean Difference (Net) = 3.4, 90% CI 2-sided [-0.7 to 7.6], Standard Error of Mean 2.5 — Difference = (adjusted mean 5 mg BI 1358894) - (adjusted mean Placebo)
Statistical Analysis 2: Comparison: Placebo vs 25 mg BI 1358894; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.0757, Mixed Models Analysis; Mean Difference (Net) = 4.4, 90% CI 2-sided [0.3 to 8.5], Standard Error of Mean 2.5 — Difference = (adjusted mean 25 mg BI 1358894) - (adjusted mean Placebo)
Statistical Analysis 3: Comparison: Placebo vs 75 mg BI 1358894; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.6864, Mixed Models Analysis; Mean Difference (Net) = 1.0, 90% CI 2-sided [-3.0 to 5.0], Standard Error of Mean 2.4 — Difference = (adjusted mean 75 mg BI 1358894) - (adjusted mean Placebo)
Statistical Analysis 4: Comparison: Placebo vs 125 mg BI 1358894; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.1585, Mixed Models Analysis; Mean Difference (Net) = 2.8, 90% CI 2-sided [-0.5 to 6.0], Standard Error of Mean 1.9 — Difference = (adjusted mean 125 mg BI 1358894) - (adjusted mean Placebo)

ADVERSE EVENTS:
Time Frame: From first treatment administration until last treatment administration + 28 days, up to approximately 11 weeks.
Description: Treated Set (TS): all participants that have been randomized and that received at least one administration of study drug. Participants are analysed according to the actual received treatment.
Arm/Group | Placebo | 5 mg BI 1358894 | 25 mg BI 1358894 | 75 mg BI 1358894 | 125 mg BI 1358894 | Quetiapine
All-Cause Mortality (participants affected / at risk) | 0/128 | 0/36 | 0/39 | 0/39 | 0/75 | 0/71
Serious Adverse Events (participants affected / at risk) | 7/128 | 0/36 | 2/39 | 2/39 | 1/75 | 1/71
Other Adverse Events (participants affected / at risk) | 32/128 | 16/36 | 22/39 | 24/39 | 34/75 | 43/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=128) | 5 mg BI 1358894 (N=36) | 25 mg BI 1358894 (N=39) | 75 mg BI 1358894 (N=39) | 125 mg BI 1358894 (N=75) | Quetiapine (N=71)
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Emotional distress (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 6 | 0 | 0 | 2 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=128) | 5 mg BI 1358894 (N=36) | 25 mg BI 1358894 (N=39) | 75 mg BI 1358894 (N=39) | 125 mg BI 1358894 (N=75) | Quetiapine (N=71)
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 2 | 0 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 4 | 0 | 2 | 1 | 1 | 4
Fatigue (General disorders) | 4 | 5 | 3 | 2 | 4 | 7
COVID-19 (Infections and infestations) | 5 | 1 | 1 | 3 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2 | 2 | 2 | 3
Respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 2 | 2 | 3 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 2 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 2 | 6 | 2 | 4 | 6
Headache (Nervous system disorders) | 13 | 9 | 4 | 4 | 13 | 2
Sedation (Nervous system disorders) | 1 | 0 | 1 | 2 | 2 | 6
Somnolence (Nervous system disorders) | 4 | 1 | 1 | 7 | 5 | 24
Aggression (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 0 | 0 | 2 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 2 | 1 | 2 | 6
Sleep disorder (Psychiatric disorders) | 2 | 0 | 2 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT04521478/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT04521478/SAP_001.pdf